CLINICAL TRIAL: NCT00986843
Title: A Phase I Clinical Trial to Determine the Maximum Tolerated Dose and to Assess the Safety and Pharmacokinetic Profile of OratecanTM in Patients With Advanced Solid Cancer((Q1DX5/W)X2 for 3W)
Brief Title: Clinical Trial to Evaluate Safety and Tolerability of OratecanTM in Patients With Advanced Solid Malignancies (Oratecan-102)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-OTE-102
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Advanced Solid Malignancies
Keywords: HM30181A; Irinotecan; MTD; DLT
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HM30181AK tablet + Irinotecan tablets (Experimental): HM30181AK tablet + Irinotecan tablets
  Interventions: Drug: HM30181AK tablet + Irinotecan tablets

INTERVENTIONS:
Drug: HM30181AK tablet + Irinotecan tablets — HM30181AK 60 mg tablet + Irinotecan 20mg, 5 mg or 2mg tablets

SUMMARY:
The main objective of this study is to determine the maximum tolerated dose (MTD) of OratecanTM. Eligible subjects of this study are patients with histologically or cytologically confirmed malignant solid tumor refractory to standard therapy.

The irinotecan hydrochloric acid (HCl) tablet is escalated and administered per body surface area (BSA). The dose of HM30181A 60 mg is fixed.

The Route of administration of irinitecan and HM30181A is oral. Each cycle consists of 21 days. Drugs are administered daily for 10 consecutive days (D1, 2, 3, 4, 5, 8, 9, 10, 11 and 12) followed by a washout of 9 days.

DETAILED DESCRIPTION:
Besides the main objective, there are 3 other objectives as follows.

1. To determine dose-limiting toxicity (DLT) of OratecanTM
2. To characterize the pharmacokinetics of HM30181A, irinotecan and its metabolites (SN-38 and SN-38G) following oral administration of OratecanTM
3. To evaluate anticancer activity of OratecanTM in patients with advanced solid malignancies Groups of 3 patients per cohort or dose level will be treated with escalating doses of irinotecan in combination with a fixed 60mg dose of HM30181A.

If 0/3 patients at any dose level experience a DLT, the dose of irinotecan will be escalated by 10 mg/m2 in the next dose level. If 1/3 patients at any dose level experience a DLT, the cohort will be expanded by 3 additional patients to 6 patients. If no additional patients develop DLT, the dose of irinotecan will again be escalated in the next cohort of 3 patients. If 2/3 or 2/6 patients develop DLT, then dose escalation will cease, and the previous dose will be declared the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumors
* Patients who have experienced progressive disease despite of conventional anticancer therapy. Patients who cannot expect effective treatment or prolonged survival with conventional anticancer therapy
* Previous chemotherapy (excluding irinotecan), radiotherapy and surgical operation are allowed if they are discontinued for at least 4 weeks prior to D0 and all adverse events are resolved (6 weeks for nitrosoureas and mitomycin)
* Aged ≥18
* Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2
* A life expectancy greater than 12 weeks
* Adequate bone marrow (platelet≥100 x 109/L, hemoglobin≥10.0g/dl and ANC≥ 1.5 x 109/L, renal (Creatinine≤1.5mg/dl) and liver function (AST/ALT/ALP ≤ 3 x upper limit of normal and total bilirubin≤2mg/dl) and no abnormal heart and lung function However, AST/ALT/ALP ≤ 5 x upper limit of normal for patients with liver metastases and ALP level ≤ 5 x upper limit of normal for patients with bone metastases are allowed.
* Patients with no need of radiotherapy (except for true oncologic emergency occurring after entry on study [e.g. acute spinal cord compression], other anticancer drugs and immunotherapy during the trial
* Subjects must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up assessments and procedures

Exclusion Criteria:

* Patients with hematopoietic malignancies ( including leukemia, lymphoma, multiple myeloma, myelodysplastic syndromes, myeloproliferative disorders), ileus, CNS metastasis, and with active infections requiring parenteral or systemic antibacterial, antiviral, or antifungal therapy. Patients with infections may participate in this clinical trial after complete recovery or control of the infection
* Patients with chronic malabsorption, or who have undergone total colectomy
* Patients who have undergone hematopoietic stem cell transplantation (HSCT) or are candidates for planned HSCT
* History of congestive heart failure, atrial arrhythmia or ventricular arrhythmia requiring medication; Patients who had treatment for myocardial infarction or any other acute coronary syndrome event within the past 6 months.
* Subjects who, in the investigator's opinion, cannot be treated per protocol due to functional impairments due to any other severe co-morbid medical conditions
* Pregnant or breast-feeding patients; Women of childbearing potential without adequate contraception (Men must use adequate contraception.)
* Subjects who have no intention of following the requirements of the protocol or the follow-up management. Subjects who cannot be followed up regularly due to psychological, social, family, logistic, and geographical reasons.
* Subjects who have been treated with PGP inhibitors (cyclosporine A and verapamil), which are contraindicated medications, will have a wash-out period of 2 weeks.
* Subjects who were administered with other investigational products within 28 days before screening.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Toxicity evaluation (safety evaluation): Toxicity will be evaluated by medical history, vital signs, physical examination and laboratory tests performed during the screening period (D-28 to D0) and treatment period based on NCI-CTCAE (version 3.0). | Toxicity will be evaluated on Day 21 during Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yoo Kim, M.D. Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea